CLINICAL TRIAL: NCT00385125
Title: Phase II Study for Treatment of Patients With Relapsed or Primary Refractory Aggressive B- Cell NHL and Anthracycline Chemotherapy Pretreatment, Who Received or Did Not Qualify for Autologous Stem Cell Transplantation.
Brief Title: Treatment of Patients With Relapsed or Primary Refractory Aggressive B- Cell NHL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Magdeburg (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSHO #73
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2006-10

CONDITIONS: Lymphoma, High-Grade
Keywords: relapsed; refractory; CD 20 positive
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — Bendamustine Hydrochloride; Rituximab

INTERVENTIONS:
Drug: Bendamustine
Drug: Rituximab

SUMMARY:
Phase II study for treatment of patients with relapsed or primary refractory aggressive B- cell NHL and anthracycline chemotherapy pretreatment, who received or did not qualify for autologous stem cell transplantation.

DETAILED DESCRIPTION:
Phase II study for treatment of patients with relapsed or primary refractory aggressive B- cell NHL and anthracycline chemotherapy pretreatment, who received or did not qualify for autologous stem cell transplantation. Aim is to find response rates and duration of combination chemotherapy (bendamustine/rituximab) in patients with relapsed or refractory CD 20 positive B cell NHL.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven high grade B-NHL (CD 20 >= 20 % positive)
* Age >= 18 years
* At least one pretreatment with anthracycline polychemotherapy +/- radiatio:
* first relapse nad contraindication for aggressive salvage therapy e.g. high dose therapy with autologous stem cell transplantation
* second relapse (after aggressive salvage therapy)
* patient's refusal of aggressive salvage therapy in first relapse
* informed consent

Exclusion Criteria:

* untreated patients
* pretreatment with bendamustine
* primary CNS- lymphoma
* Karnofsky index < 50 (except caused by lymphoma)
* HIV positive, hepatitis B or C
* serious concurrent disease
* non-compensated heart failure (>=NYHA 3)
* non-compensated hypertension
* renal insufficiency (creatinine > 2.0 mg/dl), not related to lymphoma
* hepatic insufficiency with transaminase values greater than 3-fold of normal values and/or bilirubin levels > 200 µmol/l, not related to lymphoma
* missing compliance respective incapability to comply (e.g.cerebral dysfunction
* pregnancy
* hematopoetic insufficiency not lymphoma related (leucocyte count <= 2500/µl, granulocyte count <= 1000/µl, platelet count <= 80000/µl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-08; Study Completion 2010-08

PRIMARY OUTCOMES:
response rate
response duration

SECONDARY OUTCOMES:
overall survival
toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Martin Mohren, PD, Principal Investigator — University of Magdeburg, Department of Hematology and Oncology
Locations (1):
- University of Magdeburg, departement of Hematology and Oncology, Magdeburg, Germany